CLINICAL TRIAL: NCT02917694
Title: A Feasibility Study to Assess Pre Admission Status and Six Month Outcomes of Major Trauma Patients Admitted to an Intensive Care Unit, Using the WHO DAS 2.0.
Brief Title: A Feasibility Study to Assess Pre Admission Status and Six Month Outcomes After Major Trauma
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Rebekah Haylett, Physiotherapist, Oxford University Hospitals NHS Trust
Other Study IDs: 209899
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Multiple Trauma
MeSH Terms: conditions — Multiple Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to assess the feasibility of obtaining details about a patients previous level of function from the patient of friend/relative, after they have been admitted an intensive care unit (ICU). It will also assess the feasibility of re-assessing level of function at 6 months after the patient has been discharged from ICU.

DETAILED DESCRIPTION:
Currently there is no standardised way of obtaining details about a patients pre-admission level of function. the process of gaining this history is often done by several different people with no standard questions asked.

There is also a need to be able to measure what happens to patients after they leave ICU, and compare their abilities to preadmission status.

This feasibility study will aim to investigate:

* the time taken to train the physiotherapy team in the use of the outcome measure
* the ability to obtain pre admission functional status from patients/friend/relative on admission to ICU
* the ability to follow patients up at 6 months post discharge with re-assessment of the outcome measure

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Participants relative or friend (consultee) is willing and able to give informed consent for participation in the study (where the patient is unable to give informed consent)
* Male or Female, aged 18 years or above
* Injury Severity Score greater than 9
* Admitted as an emergency to AICU
* Experienced at least 24 hours level three care during their admission

Exclusion Criteria:

* Non UK resident (due to potential loss to follow up)
* Unwilling to consent
* No GP details available
* Patients with a palliative diagnosis or established on a palliative treatment pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU after multiple trauma
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
WHODAS 2.0 completion rate | 2 days
  Number of questionnaires completed/returned on admission to ICU

SECONDARY OUTCOMES:
Time to questionnaire completion rate | 2 days
  The time taken (hours) from ICU admission to complete the questionnaire
WHODAS 2.0 completion rate | 6 months post ICU discharge
  Number of questionnaires completed/returned at 6 months post ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah Haylett, BSc (Hons), Principal Investigator — Oxfod University Hospitals NHS Foundation Trust
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No